CLINICAL TRIAL: NCT03621592
Title: An Exploratory, Single Center, Observer Masked, Active Control, Randomized Trial to Investigate the Effectiveness of Dialkylcarbomoyl Chloride Dressing (Cutimed Sorbact) in Modifying Bacterial Load in Venous Leg Ulcers (VLU)
Brief Title: VLU Dressing Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: BSN Medical Inc (Industry)
Responsible Party: Principal Investigator, Hadar Lev-Tov, Assistant professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20180468
Record Dates: First submitted 2018-07-20; First posted 2018-08-08 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study and products, investigator blinding is unrealistic and subject blinding is unlikely. Research staff will avoid naming the dressing or suggesting the assignment to the subjects. However, an independent monitor with experience in treating wounds will be blinded to the treatment assignment and will confirm healing outcomes based on images.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cutimed® Sorbact® (Experimental): Participants in this group will receive the Cutimed Sorbact intervention for 6 weeks.
  Interventions: Device: Cutimed® Sorbact®
- Acticoat® (Active Comparator): Participants in this group will receive the Acticoat intervention for 6 weeks.
  Interventions: Device: Acticoat®

INTERVENTIONS:
Device: Cutimed® Sorbact® — Dialkylcarbomoyl chloride based wound dressing
  Arms: Cutimed® Sorbact®
Device: Acticoat® — Silver impregnated contact layer dressing
  Arms: Acticoat®

SUMMARY:
The goal of the study is to investigate the effectiveness of Cutimed Sorbact (Study Device) in modifying bacterial load in venous leg ulcers (VLU).

ELIGIBILITY:
Inclusion Criteria:

1. Adults, 18 years old and older (i.e. age ≥ 18 years).
2. Venous leg ulcer (VLU) is present on the leg. VLU shall be full thickness but without exposure of deeper tissues (muscle bone or tendon).
3. If more than one ulcer is present, the largest ulcer meeting criteria shall be designated the study ulcer.
4. If more than one ulcer on the study ulcer limb, study ulcer shall be at least one centimeter from other ulcers.
5. Venous Doppler ultrasound exam, within one year from randomization, shall demonstrate reflux of over 0.5 seconds in the affected limb.
6. Ankle-Brachial Pressure Index (ABI) exam with value of ≥0.80 in the affected limb
7. VLU has been treated with silver based therapy for at least 2 weeks within the previous 6 months.
8. VLU present for at least one month prior to screening visit 1.
9. VLU at least 2 cm2 in size but not larger than 100 cm2.
10. After debridement, study ulcer demonstrates a clean wound bed.
11. If subject is a female of childbearing potential, subject must use at least one method of contraception acceptable by PI such as birth control pills, Intrauterine Device (IUD), condoms, or sexual abstinence. At visit 1 urine pregnancy test must be negative.
12. Subject is able to comprehend all study related procedures and adhere to study schedule.
13. Subject is able to provide written informed consent.

Exclusion Criteria:

1. Based on investigator medical judgment, ulcer is caused by any etiology exclusive of venous insufficiency.
2. Study Ulcer surface area (post-debridement) has increased or decreased by more than 30% in the period between screening visit 1 and treatment visit 1.
3. Study Ulcer exhibits clinical signs and symptoms of infection in the period between screening visit 1 and treatment visit 1 requiring oral antibacterial therapy.
4. Subject has known allergy to any of the materials used in the study.
5. Subject is unable to tolerate multi-layer compression therapy.
6. Based on investigator medical judgment, the Study Ulcer is suspicious for cancer (e.g. basal cell carcinoma or squamous cell carcinoma).
7. In the month prior to screening visit 1 subject was treated with systemic immunosuppressive medications for more than 2 weeks (e.g. chemotherapy, corticosteroids), and/or it is anticipated subject will require such medications during study period.
8. In the month prior to screening visit 1 subject was enrolled in any other research protocol for treatment of Study Ulcer.
9. The Subject has been diagnosed with malignant disease not in remission over the 5 years immediately preceding screening visit 1. (Except: cervical carcinoma in situ, cutaneous squamous cell carcinoma, cutaneous basal cell carcinoma that have been treated and have no evidence of recurrence or metastases).
10. Study ulcer area has been treated with radiation therapy at any time.
11. In the opinion of PI the subject has a medical condition such as autoimmune, renal, hepatic or hematologic disease that makes the subject an inappropriate candidate for participation in study.
12. In the month preceding screening visit 1 Study Ulcer has been treated with advanced tissue engineered devices matrix based devices (e.g., Apligraf, Dermagraft, Oasis).
13. Subject is diagnosed with New York Heart Association Class III and IV congestive heart.
14. Failure: Class III: Symptoms with moderate exertion or, Class IV: Symptoms at rest.
15. Subject is diagnosed with diabetes mellitus that is poorly controlled and shall be defined as hemoglobin A1C >10%.
16. Study Ulcer is completely or more than 50% of the Study Ulcer is located on the foot (i.e. below the malleolus).
17. Subject is a female of childbearing potential, and refusing to use at least one method of contraception acceptable by PI such as birth control pills, IUD, condoms, or sexual abstinence.
18. Positive pregnancy test in screening visit 1 in a female of childbearing potential or active pregnancy or breast-feeding.
19. In the opinion of the PI the subject is unable to understand or comply with study related protocol including but not limited to providing informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hadar Lev-Tov, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cutimed® Sorbact® | Acticoat®
Started | 15 | 16
Completed | 12 | 14
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Lack of Improvement | 1 | 0
Not completed — Preference to receive wound care closer to home | 1 | 0
Not completed — Lack of healing | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cutimed® Sorbact® | Acticoat® | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 12 | 22
  >=65 years | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.33 (12.81) | 58.25 (10.44) | 58.77 (11.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 8 | 9 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 5 | 14
  Not Hispanic or Latino | 6 | 11 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 9 | 10 | 19
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Childbearing potential [Count of Participants; unit: Participants] | 1 | 0 | 1
Weight [Mean (Standard Deviation); unit: kilograms] | 90.84 (20.73) | 97.93 (21.68) | 94.12 (20.64)
Height [Mean (Standard Deviation); unit: centimeters] | 173.44 (11.80) | 172.93 (10.95) | 173.0 (11.19)
Tobacco use [Count of Participants; unit: Participants] | 15 | 16 | 31
Length of tobacco use [Mean (Standard Deviation); unit: years (mean)] — Length of tobacco use in years (mean)
  years (mean) | 26.5 (13.43) | 24.69 (16.48) | 25.29 (14.29)
Tobacco cessation years [Mean (Standard Deviation); unit: years] | 23 (17.3) | 12 (4.24) | 17.5 (10.77)

OUTCOME MEASURES:

1. Primary Outcome: Change in Bacterial Load
Description: Mean change in bacterial load in Colony Forming Units (CFU)/grams will be assessed from tissue samples
Time Frame: Baseline, Up to 8 weeks
Measure: Mean (Standard Deviation); unit: CFU/gram
Arm/Group | Cutimed® Sorbact® | Acticoat®
Number analyzed (Participants) | 11 | 12
CFU/gram | 12678.81 (23698.6) | 33190.8 (57882.61)

2. Secondary Outcome: Wound Healing Rate
Description: Wound healing rate (in cm^2/week) will be calculated by measuring the wound area
Time Frame: Up 6 weeks
Measure: Mean (Standard Deviation); unit: cm^2/week
Arm/Group | Cutimed® Sorbact® | Acticoat®
Number analyzed (Participants) | 15 | 16
cm^2/week | .179 (.272) | .122 (.258)

3. Secondary Outcome: Percentage of Subjects With Complete Healing
Description: The percentage of subjects achieving complete healing of ulcer at the evaluation of treating physician will be reported
Time Frame: Up to 8 weeks
Measure: Number; unit: percent of patients
Arm/Group | Cutimed® Sorbact® | Acticoat®
Number analyzed (Participants) | 15 | 16
percent of patients | 20 | 0

4. Secondary Outcome: Pain as Measured by VAS Scores
Description: The Pain Visual Analog Scale (VAS) has range from 0 (no pain) to 100 (worst possible pain). Mean change in scores will be reported from last visit compared to baseline will be reported.
Time Frame: Up to 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cutimed® Sorbact® | Acticoat®
Number analyzed (Participants) | 7 | 8
units on a scale | .43 (34.9) | -16.9 (18.9)

5. Secondary Outcome: Wound Quality of Life (WQoL) Scores
Description: WQoL is a 17 item questionnaire with each question scored on a 5 point scale, where 0 is "not at all" and 5 is "very much". WQoL has a total score ranging from 0 to 85 with a lower score indicating better quality of life. Mean change in scores will be reported from last visit compared to baseline will be reported.
Time Frame: Up to 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cutimed® Sorbact® | Acticoat®
Number analyzed (Participants) | 11 | 14
units on a scale | -9.1 (14.5) | -4.1 (11.1)

6. Secondary Outcome: EQ-5D-5L Quality of Life Scores
Description: The Euro Quality of life-5-Dimension-5-Level (EQ-5D-5L) is averaged based off the 5 point scale, where 0 is "no problems" and 5 is "extreme problems". Difference in scores will be reported from last visit compared to baseline will be reported.
Time Frame: Up to 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cutimed® Sorbact® | Acticoat®
Number analyzed (Participants) | 12 | 14
units on a scale | 0.12 (0.23) | 0.08 (0.13)

7. Secondary Outcome: Number of Adverse Events
Description: As assessed by treating physician
Time Frame: Up to 8 weeks
Measure: Number; unit: number of adverse events
Arm/Group | Cutimed® Sorbact® | Acticoat®
Number analyzed (Participants) | 15 | 16
number of adverse events | 3 | 2

ADVERSE EVENTS:
Time Frame: Up to 8 weeks from start date
Arm/Group | Cutimed® Sorbact® | Acticoat®
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 3/15 | 2/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cutimed® Sorbact® (N=15) | Acticoat® (N=16)
Cutaneous infection (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Squamous cell carcinoma

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-17): https://cdn.clinicaltrials.gov/large-docs/92/NCT03621592/Prot_SAP_000.pdf